CLINICAL TRIAL: NCT05614232
Title: Single-Center, Retrospective, Pivotal Study to Evaluate the Effectiveness of Investigational Device (Lunit INSIGHT CXR) in Detection of Abnormal Findings on Chest Radiographs
Brief Title: Study to Evaluate the Effectiveness of the Device in Detection of Abnormal Findings on Chest X-ray
Status: Completed | Type: Observational
Sponsor: Lunit Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LUN_CXR_CA_221
Record Dates: First submitted 2022-11-02; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive group: chest radiographs with the specific target radiologic findings (Atelectasis, Calcification, Cardiomegaly, Consolidation, Fibrosis, Mediastinal Widening, Nodule/Mass, Pleural Effusion, Pneumoperitoneum, Pneumothorax)
  Interventions: Radiation: Chest X-ray
- Negative group: chest radiographs with no target radiologic findings
  Interventions: Radiation: Chest X-ray

INTERVENTIONS:
Radiation: Chest X-ray — Chest radiographs

SUMMARY:
This study aims to evaluate the effectiveness of the investigational device (Lunit INSIGHT CXR) in the detection of chest abnormalities

DETAILED DESCRIPTION:
In the study, the standalone performance of Lunit INSIGHT CXR was primarily assessed by comparing the analysis results from the investigational device and reference standards in the detection of 10 abnormal radiologic findings - atelectasis, calcification, cardiomegaly, consolidation, fibrosis, mediastinal widening, nodule/mass, pleural effusion, pneumoperitoneum, and pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiographs of aged 14 years or older
* Conventional PA or AP chest radiographs
* Chest radiographs with confirmed radiology reports

Exclusion Criteria:

* Chest radiographs taken in postures other than PA and AP
* Chest radiographs from dual-energy radiography
* Invert-grayscale chest radiographs

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Secondary hospital patient
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
the effectiveness of the investigational device | through study completion, an average of 6 months
  Area Under the Receiver Operating Characteristic Curve (ROC AUC) of the investigational device in detection of overall target radiologic findings (detection of any abnormal findings among ten target radiologic findings)

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No